CLINICAL TRIAL: NCT04417205
Title: Isolating and Exploiting the Mechanisms That Link Breakfast and Human Health - Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, James Betts, Professor James Betts, University of Bath
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: DC-I
Record Dates: First submitted 2019-03-05; First posted 2020-06-04 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Physical Activity; Postprandial Metabolism; Weight Loss
MeSH Terms: conditions — Motor Activity; Weight Loss

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to one of 3 intervention arms.
Who Masked: Participant
Masking Description: Where applicable (i.e. the two breakfast feeding interventions) participants will be blinded to the breakfast that they receive for 28-days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Carbohydrate rich breakfast (Active Comparator): Participants will be provided with 28-days worth of pre-weighed carbohydrate rich breakfast materials to consume before 1000h daily.
  Interventions: Other: Carbohydrate Rich Breakfast
- Whey protein enriched breakfast (Experimental): Participants will be provided with 28-days worth of pre-weighed whey protein enriched rich breakfast materials to consume before 1000h daily.
  Interventions: Dietary Supplement: Whey protein enriched breakfast
- Extended morning fast (No Intervention): Participants will be asked to remain fasted (i.e. to not consume breakfast) until 1200h daily for 28-days.

INTERVENTIONS:
Other: Carbohydrate Rich Breakfast — Participants will be asked to consume the provided carbohydrate rich breakfast before 1000h daily for 28 days.
  Arms: Carbohydrate rich breakfast
Dietary Supplement: Whey protein enriched breakfast — Participants will be asked to consume the provided whey protein enriched breakfast before 1000h daily for 28 days.
  Arms: Whey protein enriched breakfast

SUMMARY:
Following the establishment of causal links between breakfast consumption, the individual components of energy balance, and health it is now important to examine and target the underlying biological mechanisms involved to maximise potential health benefits.

To begin investigating the outlined mechanisms healthy, non-obese participants will be recruited to take part in phase I (acute design) of a wider project.

DETAILED DESCRIPTION:
Causal links between breakfast consumption, the individual components of energy balance, and health have recently been established and it is now important to examine and target the underlying biological mechanisms over a longer period of time to maximise potential health benefits.

Specifically, the substitution of a portion of carbohydrate for protein at breakfast may enhance the potential health benefits of breakfast through targeting distinct mechanistic pathways. Broadly, introducing a greater protein load at breakfast increases insulin secretion and delays gastric emptying, thereby eliciting a potentiated insulin response. In turn this may therefore improve glucose tolerance during a subsequent meal. Additionally, maintenance of euglycaemia following breakfast consumption, coupled with the thermic effect of feeding protein may accentuate the elevated energy expenditure following breakfast observed in previous studies. Finally, both the physical and chemical properties of protein exert a marked satiating effect. Collectively, these mechanisms could interact to maximise the net impact of breakfast on energy balance and associated health outcomes. However, whilst the evidence indicates obvious benefits of feeding a higher protein dose at breakfast, relatively little research has focused on the response to protein over multiple meals/days. Furthermore, and importantly, the mechanisms involved in the second-meal phenomenon and the potential for initial meals of varied composition to target these mechanisms have never been systematically investigated.

To begin investigating the outlined mechanisms healthy, non-obese participants will be recruited to undergo a 4 week intervention study in which they will consume one of three breakfasts for 28-days. The breakfast interventions provide will be:

Carbohydrate rich breakfast

Whey protein enriched breakfast

Extended morning fast

Participants will undergo 7 days of habitual physical activity and diet monitoring prior to visiting the laboratory for their preliminary metabolic assessment in which they will consume the carbohydrate rich breakfast followed by an ad libitum meal for lunch. They will then be randomised to one of the 3 breakfast interventions for 28-days. During the 28-days weekly monitoring of physical activity and energy intake will take place in order to assess energy balance.

Upon completion of the intervention phase participants will revisit the laboratory to replicate the initial visit in which postprandial metabolism was assessed.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 18.5-29.9 kg∙m-2
* Age 18-65 years
* Able and willing to provide informed consent and safely comply with study procedures
* Females to maintain record of regular menstrual cycle phase or contraceptive use
* No anticipated changes in diet/physical activity during the study (e.g. holidays or diet plans)
* Inclusive to all breakfast habits (e.g. regular skipper / consumer)

Exclusion Criteria:

* Any reported condition or behaviour deemed either to pose undue personal risk to the participant or introduce bias
* Any diagnosed metabolic disease (e.g. type 1 or type 2 diabetes)
* Any reported use of substances which may pose undue personal risk to the participants or introduce bias into the experiment (e.g. smoking/substance abuse)
* Lifestyle not conforming to standard sleep-wake cycle (e.g. shift worker)
* Any reported recent (<6 months) change in body mass (± 3%)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-02-26 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-08-01 (Actual)

PRIMARY OUTCOMES:
Change in physical activity thermogenesis | Assessed for 1 week at baseline, 3 days a week during weeks 1-3 of the intervention and again for 1 week in the 4th week of the intervention.
  Energy expenditure measured using physical activity monitor
Change in expression of circadian clock genes measured in whole blood | Baseline and 4-weeks
  Pre and post intervention change clock gene expression
Change in postprandial glycaemia following carbohydrate rich test breakfast and lunch over 4 weeks | Baseline and 4-weeks
  The postprandial time course response of plasma glucose to the test breakfast and lunch meals
Change in postprandial insulinaemia following carbohydrate rich test breakfast and lunch over 4 weeks | Assessed at baseline and after 4 weeks of the intervention
  The postprandial time course response of plasma insulin to the test breakfast and lunch meals
Change in body mass | 4 weeks
  Participants will be weighed prior to the intervention and again upon completion

SECONDARY OUTCOMES:
Change in postprandial incretin hormone response following breakfast and lunch | Baseline and 4 weeks
  The postprandial time course response of plasma incretin hormones (e.g. GLP-1 & GIP) to the the test breakfast.
Change in subjective appetite ratings following breakfast and lunch | Baseline and 4 weeks
  Ratings of appetite provided on subjective appetite scales (on a scale of 0-100 mm where 0 is associated with lower ratings and 100 with higher ratings) following the test breakfast and lunch
Change in fuel oxidation during the test breakfast | Baseline and 4 weeks
  Fat and carbohydrate oxidation following breakfast

CONTACTS AND LOCATIONS:
Overall Officials: Harry A Smith, MSci, Principal Investigator — University of Bath; James A Betts, PhD, Principal Investigator — University of Bath
Locations (1):
- University of Bath, Bath, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Leidy HJ, Ortinau LC, Douglas SM, Hoertel HA. Beneficial effects of a higher-protein breakfast on the appetitive, hormonal, and neural signals controlling energy intake regulation in overweight/obese, "breakfast-skipping," late-adolescent girls. Am J Clin Nutr. 2013 Apr;97(4):677-88. doi: 10.3945/ajcn.112.053116. Epub 2013 Feb 27. PMID 23446906
- [Background] Bray GA, Redman LM, de Jonge L, Covington J, Rood J, Brock C, Mancuso S, Martin CK, Smith SR. Effect of protein overfeeding on energy expenditure measured in a metabolic chamber. Am J Clin Nutr. 2015 Mar;101(3):496-505. doi: 10.3945/ajcn.114.091769. Epub 2015 Jan 14. PMID 25733634
- [Background] Park YM, Heden TD, Liu Y, Nyhoff LM, Thyfault JP, Leidy HJ, Kanaley JA. A high-protein breakfast induces greater insulin and glucose-dependent insulinotropic peptide responses to a subsequent lunch meal in individuals with type 2 diabetes. J Nutr. 2015 Mar;145(3):452-8. doi: 10.3945/jn.114.202549. Epub 2014 Dec 24. PMID 25733459
- [Background] Chowdhury EA, Richardson JD, Holman GD, Tsintzas K, Thompson D, Betts JA. The causal role of breakfast in energy balance and health: a randomized controlled trial in obese adults. Am J Clin Nutr. 2016 Mar;103(3):747-56. doi: 10.3945/ajcn.115.122044. Epub 2016 Feb 10. PMID 26864365
- [Background] Betts JA, Richardson JD, Chowdhury EA, Holman GD, Tsintzas K, Thompson D. The causal role of breakfast in energy balance and health: a randomized controlled trial in lean adults. Am J Clin Nutr. 2014 Aug;100(2):539-47. doi: 10.3945/ajcn.114.083402. Epub 2014 Jun 4. PMID 24898233